CLINICAL TRIAL: NCT04134585
Title: Promoting Fall Prevention Workshops for Individuals Aged 60 and Over: an Exploratory Study.
Brief Title: Promoting Fall Prevention Workshops
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Crédit Agricole Loire / Haute-Loire (Unknown); Jean Monnet University (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN912018/CHUSTE
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Behavior; Aging
Keywords: Fall; Prevention; Seniors; Physical activity; Interviews
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People aged 60: People aged 60 and over who had refused to participate in fall prevention workshops will be included. They will have semi-structured interviews.
  Interventions: Other: semi-structured interviews

INTERVENTIONS:
Other: semi-structured interviews — Semi-structured interviews will be performed to determine representations of physical activity, reluctance/motivation to participate in physical activity sessions and facilitators who can help them overcome these barriers.

SUMMARY:
Physical Activity (PA) is recognized as the most effective method to prevent falls in the elderly. Yet despite there being a consensus now that Physical Activity (PA) is effective in practice, there remain many obstacles to participation resulting in PA approaches designed to prevent falls actually only benefiting a limited number of elderly subjects.

DETAILED DESCRIPTION:
It's a qualitative study. The target population was people aged 60 and over who had refused to participate in fall prevention workshops.

The study covered three different French departments. A total of 19 semi-structured interviews were conducted over a period of 5 months.

The analysis of reports revealed there were multiple motives for not participating in the balance workshops. The current means of promoting these fall prevention workshops are not adapted. Finally, the social experience provided by the program was identified to be the principal motivator for encouraging the interviewed subjects to participate.

ELIGIBILITY:
Inclusion Criteria:

* People who received a proposal to participate in our workshop and who denied it
* People living in one of the three departments of the study (Loire, Haute-Loire and Rhône)

Exclusion Criteria:

- People who refused to participate to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People aged 60 and over.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Correlation between physical activity degree, aging and illness | Month: 5
  Analysis interview responses.

SECONDARY OUTCOMES:
Analysis representations of physical activity. | Month: 5
  Analysis interview responses.
Analysis reluctance to participate in physical activity sessions. | Month: 5
  Analysis interview responses.
Analysis motivation to participate in physical activity sessions. | Month: 5
  Analysis interview responses.
Analysis facilitators who can help them overcome these barriers | Month: 5
  Analysis interview responses.

CONTACTS AND LOCATIONS:
Overall Officials: Luc GOETHALS, Doctoral student, Principal Investigator — Jean Monnet University
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No